CLINICAL TRIAL: NCT03265834
Title: The CABI Trial: An Unblinded Parallel Group Randomised Controlled Feasibility Trial of Long Course Antibiotic Therapy (28 Days) Compared to Short Course (≤10 Days) in the Prevention of Complicated Intra-ABdominal Infection Relapses in Adults Treated for Complicated Intra-ABdominal Infection
Brief Title: CABI: Antibiotic Duration for Complicated Intra-ABdominal Infection
Acronym: CABI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Andrew Kirby, Associate clinical professor, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MB16/156
Record Dates: First submitted 2017-08-23; First posted 2017-08-29 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Complicated Intraabdominal Infections
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Long course antibiotic therapy (28 days) (Experimental): Antibiotic therapy for a duration of 28 days
  Interventions: Other: 28 days of antibiotics
- Short course antibiotic therapy (≤10 days) (Active Comparator): Antibiotic therapy for a duration of ≤10 days
  Interventions: Other: < 10 days of antibiotics

INTERVENTIONS:
Other: < 10 days of antibiotics — Antibiotic duration
  Arms: Short course antibiotic therapy (≤10 days)
Other: 28 days of antibiotics — Antibiotic duration
  Arms: Long course antibiotic therapy (28 days)

SUMMARY:
Complicated intra-ABdominal Infections (CABIs) are abdominal infections where there is an abscess inside the abdomen, or a hole (perforation) in an abdominal organ such that infected material e.g. faeces, leaks into the abdominal cavity. A recent review of CABIs after gut surgery found that they can occur in several ways. They can occur in different parts of the abdomen, can be different sizes, and may or may not be caused by a perforated bowel. Management includes, where possible, surgical drainage of an abscess or treatment of the damaged bowel. In addition, all patients are given antibiotic therapy. Despite the varied ways that CABIs occur, we currently tend to treat all CABIs with antibiotics in a similar way. CABIs are associated with significant morbidity and mortality. Despite a significant amount of disease there is little clinical evidence with which to base treatment on. One research study evaluated a short course of antibiotics (4 days) compared with a longer course (up to 10 days) in combination with surgical removal of infection. There was little difference in outcomes, but in both groups about 1 out of every 7 patients had a relapse. A recent review of patients with CABI in Leeds, not in a research study and where surgical removal infection is uncommon and antibiotic durations were short, showed that the risk of relapse was even higher (about 1 in every 3 patients). The antibiotic management of CABIs in the UK is variable and involves giving between 4 days to 28 days of antibiotics.

In summary, there is an unacceptably high relapse rate in patients treated for CABI, and uncertainty about the best length of antibiotic therapy that should be used to prevent these relapses. We therefore propose to investigate if long course antibiotic therapy (28 days) is more effective than short course antibiotics (≤10 days) in preventing relapses of CABI.

DETAILED DESCRIPTION:
Complicated intra-abdominal infection (CABI) extends beyond the hollow viscus of origin into the peritoneal space and is associated with either abscess formation or peritonitis [Solomkin 2010]. CABIs are heterogeneous in aetiology and include spontaneous infections arising from a perforated viscus, including the stomach, biliary tree, colon, appendix and reproductive organs. In addition there are post-operative complications such as peritonitis, abscess, and failure of surgical anastomoses. CABIs are also heterogeneous in their characteristics. A recent review of organ space Surgical Site Infections (SSI-Os) after colorectal surgery demonstrated that infections were varied with regard their location, as well as size and number and nature of collections, and presence of an ongoing source e.g. anastomotic breakdown (Rothwell 2016). Despite the varied origin of these infections, there are similar management strategies which centre on the source control, e.g. drainage of intra-abdominal fluid collections, and administration of antibiotic therapy. CABIs are a common in-hospital clinical challenge, in part due to the varied pathology they are caused by, and are associated with significant morbidity and mortality (DeFrances 2005, Brun-Buisson 1995). Despite this burden of disease, there is little clinical evidence with which to base treatment on, even before taking account of their heterogeneous nature. One study of CABI following source control procedures evaluated a short course of antibiotics (4 days) compared to a course of up to 2 weeks after clinical and biochemical improvement (up to 10 days). Whilst there was little difference in outcomes, both groups had a high relapse rate of approximately 15%. In addition, it is common for source control procedures not to be completed in routine clinical practice, being completed in only 17% of Leeds patients with post-operative CABI (Rothwell 2016). In this Leeds data of post-operative CABIs, where source control rates are low relapse rates were 40% (Rothwell 2016). For CABI infections, standard UK management is variable and involves between 4 and 42 days' antibiotics. This indicates an unacceptably high relapse rate in patients treated for CABI where source control is and is not undertaken. We therefore propose to investigate if long course antibiotic therapy (28 days) is clinically more effective than short course antibiotics (4 days) in preventing relapses of CABI. This study will include patients who have and have not undergone source control procedures which will be completed as per standard practice.

Complicated intra-abdominal infections require source control when possible, e.g. a surgical procedure to remove an infection, and antibiotic therapy to obtain cure. Source control is not always possible. CABIs are associated with mortality and prolongation of hospitalisation. After apparently effective treatment, potentially including source control procedures and antibiotics, infections can relapse. There are a number of reasons for relapse; one is that antibiotic treatment may not have been given for long enough to eradicate the bacteria from, what should be, a sterile intra-abdominal cavity. Antibiotics are given until a patient is better, but not until all bacteria are eradicated, allowing them to regrow and re-start an infection. Standard antibiotic duration is variable: some doctors provide long courses and others short. We therefore want to compare durations, to see if longer courses of antibiotics are able to help prevent these relapses, or if shorter courses are as effective but have fewer side effects. We have not identified closely related strategies which may optimise the management of CABIs.

The research hypothesis is therefore: In patients with CABI, regardless of source control intervention, there will be a lower relapse rate when treated with 28 days of antibiotics compared to ≤10 days of antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years
* The diagnosis of a definite CABI
* Capable of giving informed consent
* No practical or clinical barriers to consuming 28 days of antibiotic therapy, which may include consumption of antibiotics at home

Exclusion Criteria:

* a CABI diagnosed within the previous year
* a CABI diagnosed >6 days prior to screening
* uncomplicated cholecystitis/cholangitis/gall bladder empyema (no perforation or extra-biliary abscess
* a skin and soft tissue infection/abscess not communicating with the peritoneal space
* primary complicated or uncomplicated appendicitis managed surgically
* intra-abdominal infection associated with pancreatitis, pelvic inflammatory disease, primary (spontaneous) bacterial peritonitis (SBP), continuous ambulatory peritoneal dialysis peritonitis (CAPD peritonitis) and Clostridium difficile infection. concurrent infection requiring more than 10 days of therapy
* Infection with a highly resistant bacterium such that antibiotic treatment is considered to be a significantly sub-optimal by the treating microbiologist e.g. multi-resistant carbapenemase producing Entrobacteriacea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Number of participants willing to be randomised, the willingness of clinicians to allow participants to be recruited & follow up rates. | 90 days
  Screening logs, recruitment rates and follow up rates will be recorded to determine the feasibility of performing a larger study.
Number of participants who have their antibiotic therapy changed as a consequence of allocation to a certain treatment arm. | Either ≤ 10 days or 28 days depending on allocation.
  Antibiotic therapy received including any changes to treatment will be recorded.

SECONDARY OUTCOMES:
The number of participants who relapse after treatment of complicated intra-abdominal infection. | 90 days
  Frequency of complicated intra-abdominal infection (CABI) relapse with 90 days. A relapse can only occur after surgical and antibiotic therapy to manage the primary CABI has been considered successful. This will normally be demonstrated by antibiotics being stopped and no further source control procedures planned. The diagnosis of a definite CABI relapse defined as 'a combination of radiological AND clinical features consistent with CABI including a fluid collection, a temperature of ≥38 degrees and a neutrophilia (neutrophil count > 7.5 x 10*9/L) or Intra-operative confirmation of an abscess'. The diagnosis of a probable CABI relapse will be defined as ' in the absence of radiological imaging, but where no other source of infection was identified, and the patient was managed for a relapsed CABI'
Number of all infections after treatment of complicated intra-abdominal infection | 90 days
  The diagnosis of hospital acquired infections will be based on either a clinical diagnosis based on physician assessment or on definitions outlined by the 'Point prevalence survey of healthcare-associated infections and antimicrobial use in European acute-care hospitals' https://www.gov.uk/government/uploads/system/uploads/attachment_data/file/542039/ECDC_PHE_HAI_AU_PPS_2016_single_codebook.pdf
Total antibiotic consumption | 90 days
  Days of antibiotic therapy within 90 days of antibiotic therapy
Length of hospital stay within 90 days of diagnosis | 90 days
  The length of hospital stay after diagnosis of complicated intra-abdominal infection
Mortality rate after treatment of complicated intra-abdominal infection. | 90 days
  Assessed by the 90 day mortality after diagnosis of a complicated intra-abdominal infection.
The number of participants with complications from antibiotic therapy including Clostridium difficile infection (CDI) diarrhoea and catheter related blood stream infection (CRBSI) | 90 days
  Measured by the rate of adverse events, CDI and CRBSI within 90 days of diagnosis.
The number of source control procedures required for the management of CABI | 90 days
  Measured by the number source control procedures required for the management of CABI within 90 days of CABI diagnosis.
Quality of life after treatment of complicated intra-abdominal infection | Baseline, at 30 days, at 90 days and (if occurs) at time of relapse
  Assessed by a quality of life questionnaire (EQ-5D)
Feasibility of using scoring systems in complicated intra-abdominal infections | 90 days
  Measured by the ability to gather the data required to complete severity scores

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kirby, MBChB, Principal Investigator — Leeds Teaching Hospitals NHS Trust
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Solomkin JS, Mazuski JE, Bradley JS, Rodvold KA, Goldstein EJ, Baron EJ, O'Neill PJ, Chow AW, Dellinger EP, Eachempati SR, Gorbach S, Hilfiker M, May AK, Nathens AB, Sawyer RG, Bartlett JG. Diagnosis and management of complicated intra-abdominal infection in adults and children: guidelines by the Surgical Infection Society and the Infectious Diseases Society of America. Clin Infect Dis. 2010 Jan 15;50(2):133-64. doi: 10.1086/649554. PMID 20034345
- [Background] Rothwell A, Burke D, Burnside G, Kirby A. Characteristics of Organ Space Surgical Site Infection after colorectal surgery. In preparation.
- [Background] DeFrances CJ, Cullen KA, Kozak LJ. National Hospital Discharge Survey: 2005 annual summary with detailed diagnosis and procedure data. Vital Health Stat 13. 2007 Dec;(165):1-209. PMID 18350768
- [Background] Brun-Buisson C, Doyon F, Carlet J, Dellamonica P, Gouin F, Lepoutre A, Mercier JC, Offenstadt G, Regnier B. Incidence, risk factors, and outcome of severe sepsis and septic shock in adults. A multicenter prospective study in intensive care units. French ICU Group for Severe Sepsis. JAMA. 1995 Sep 27;274(12):968-74. PMID 7674528
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. Lancet. 2007 Oct 20;370(9596):1453-7. doi: 10.1016/S0140-6736(07)61602-X. PMID 18064739
- [Background] Sterne JA, White IR, Carlin JB, Spratt M, Royston P, Kenward MG, Wood AM, Carpenter JR. Multiple imputation for missing data in epidemiological and clinical research: potential and pitfalls. BMJ. 2009 Jun 29;338:b2393. doi: 10.1136/bmj.b2393. PMID 19564179
- [Background] Sawyer RG, Claridge JA, Nathens AB, Rotstein OD, Duane TM, Evans HL, Cook CH, O'Neill PJ, Mazuski JE, Askari R, Wilson MA, Napolitano LM, Namias N, Miller PR, Dellinger EP, Watson CM, Coimbra R, Dent DL, Lowry SF, Cocanour CS, West MA, Banton KL, Cheadle WG, Lipsett PA, Guidry CA, Popovsky K; STOP-IT Trial Investigators. Trial of short-course antimicrobial therapy for intraabdominal infection. N Engl J Med. 2015 May 21;372(21):1996-2005. doi: 10.1056/NEJMoa1411162. PMID 25992746
- [Derived] Ahmed S, Brown R, Pettinger R, Vargas-Palacios A, Burke D, Kirby A. The CABI Trial: an Unblinded Parallel Group Randomised Controlled Feasibility Trial of Long-Course Antibiotic Therapy (28 Days) Compared with Short Course (</= 10 Days) in the Prevention of Relapse in Adults Treated for Complicated Intra-Abdominal Infection. J Gastrointest Surg. 2021 Apr;25(4):1045-1052. doi: 10.1007/s11605-020-04545-2. Epub 2020 Mar 5. PMID 32140989

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-11-18): https://cdn.clinicaltrials.gov/large-docs/34/NCT03265834/Prot_SAP_001.pdf
  • Informed Consent Form (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT03265834/ICF_000.pdf